CLINICAL TRIAL: NCT03324269
Title: Evaluating the Predictive Value of the Nociception Level Index NOL: a Pilot Study
Brief Title: Evaluating the Predictive Value of the Nociception Level Index NOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Libre de Bruxelles (Other)
Responsible Party: Principal Investigator, Sarah Saxena, principal investigator, Université Libre de Bruxelles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NOL
Record Dates: First submitted 2017-10-16; First posted 2017-10-27 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Pain; Anesthesia
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Patients undergoing non-cardiac and cardiac surgery have NOL monitoring
Masking Description: All patients wear NOL monitoring and are aware of it. Anesthesiologist can read NOL values.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NOL (Other): After tracheal intubation and before surgical incision, a calibration Tetanus test of 100Hz, 60 mAmp during 30 sec at remifentanil level (Ce) of 4 ng/ml will be done (starting NOL below 10).
  According to the NOL response, there will be an increment of 1 ng/ml of RemiCe if NOL gradient ≥ 20 or decrement of 1 ng/ml if NOL gradient < 10. Ideal remifentanil Ce is the remifentanil Ce at which the variation of NOL index will be less than 10 units at a NOL starting value below 10. Thus this individual remifentanil Ce will be the remifentanil level programmed before surgical incision. NOL and hemodynamic responses will be recorded during the entire duration of surgery.
  Interventions: Device: NOL

INTERVENTIONS:
Device: NOL — After tracheal intubation, a Tetanus test (60 mAmp,100 Hz) is done during 30 sec at remifentanil level Ce of 4 ng/ml (with starting NOL value <10). According to the NOL response: increment of 1 ng/ml of RemiCe if NOL gradient ≥ 20 / decrement of 1 ng/ml of remifentanil Ce NOL gradient < 10. During the testing period propofol Ce is fixed at the concentration associated with BIS levels between 45-60 during the first calibration.
  Upon the incision and 2 minutes after skin incision, Propofol TCI (Schnider model) is adjusted to BIS between 45-60 and remifentanil Ce at which the variation of NOL index variation is less than10 units at a NOL starting value <10. MAP (mean arterial pressure), HR (heart rhythm) and NIBP (non-invasive blood pressure) will be measured.
  The formula derived from the calibration phase will be tested during a single tetanic stimulation at remifentanil Ce of 4 ng/ml during the validation phase.

SUMMARY:
Opioids remain the cornerstone for perioperative analgesia, albeit frequently associated with side effects. Most of these side-effects are dose-dependent.

Thus intra-operative monitors are necessary to measure the balance between Nociception and Anti-Nociception (NAN balance) by an adequate opioid administration.

Recently the NOL monitor was released.The NoL index ranges from 0 to 100 and is based on a nonlinear combination of nociception-related physiologic variables, specifically heart rate (HR), heart rate variability at the 0.15- to 0.4-Hz band power, photoplethysmograph wave amplitude (PPGA), skin conductance level, number of skin conductance fluctuations, and their time derivatives. The NoL index estimates the nociceptive/antinociceptive state from these component measures using random forest regression.

In our department, a combination of TCI propofol (Schnider model) and remifentanil (Minto model) is used to for most of the anaesthetic procedures, including cardiac anaesthesia. Remifentanil is titrated to prevent an increase in blood pressure and hearth rhythm at noxious stimuli, such as surgical incision, and adapted following hemodynamic trend during surgery.

The hypothesis of this study is to develop a calibration test using the NOL index variation to define the individual most appropriate NAN balance using remifentanil TCI before the start of surgery and before a very strong noxious surgical stimulus such as surgical incision in non-cardiac and cardiac surgery.

Before the start of surgery, the investigators want to titrate in each patient the remifentanil Ce required to abolish the NOL index response to a calibrated noxious tetanic stimulus (Tetanus 60 mamp, 100 Hz, 30 seconds). Thus this individual remifentanil Ce will be the remifentanil level programmed before surgical incision. NOL and hemodynamic responses will be recorded during the entire duration of surgery.

Study protocol amendment: validation of the calibration study: Data from the calibration phase will be used to derive a formula to predict individualised anti-nociception for incision.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing non-cardiac surgery
* Patients undergoing cardiac surgery (coronary artery bypass graft)
* Knowledge of French, English or Dutch is required.

Exclusion Criteria:

* Pregnancy
* Allergy or contraindications to one of the study drugs
* BMI >30
* History of drug and alcohol abuse,
* preoperative analgesic drug use
* Heart rhythm disturbances (Atrial fibrillation, atrial flutter).
* the use of Alpha-2 adrenergic agonists

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Predictive value of NOL | intra-operative
  A calibration Tetanus test of 60 mAmp during 30 sec at remifentanil level (Ce) of 4 ng/ml will be done when starting NOL is below 10. According to the NOL response: there will be an increment of 1 ng/ml of RemiCe if NOL gradient ≥ 10 or a decrement of 1 ng/ml of remifentanil Ce NOL gradient < 10. The optimal individual remifentanil level is defined as the level at which the variation of NOL index will be less than 10 units starting at a NOL value below 10. So surgical incision will be done at 'optimal individual remifentanil level' and MAP (mean artrial pressure), HR (heart rhythm), NIBP (non-invasive blood pressure) will be measured (every 3 minutes).

CONTACTS AND LOCATIONS:
Overall Officials: Luc Barvais, Principal Investigator — Université Libre de Bruxelles
Locations (1):
- Erasme Hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perrin L, Bisdorff M, Saxena S, Tabolcea I, Huybrechts I, Van Obbergh L, Engelman E, Barvais L, Coeckelenbergh S. Predicting personalised remifentanil effect site concentration for surgical incision using the nociception level index: A prospective calibration and validation study. Eur J Anaesthesiol. 2022 Dec 1;39(12):918-927. doi: 10.1097/EJA.0000000000001751. Epub 2022 Sep 21. PMID 36125017